CLINICAL TRIAL: NCT00377507
Title: A Clinical Trial of Tea Catechin Mouth-washing for Removal of Intraoral Bacteria in the Elderly
Brief Title: Catechin Mouth-washing for Removal of Intraoral Bacteria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult to achieve the sufficient subjects
Sponsor: Masahiro Morikawa (Other)
Responsible Party: Sponsor-Investigator, Masahiro Morikawa, Clinical trials management office, University of Shizuoka
Organization: University of Shizuoka (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT2006004
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Elderly
Keywords: catechin; elderly; mouth washing; disabled; colonized

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- catechin (Experimental): mask containing catechins
  Interventions: Dietary Supplement: catechin extracts

INTERVENTIONS:
Dietary Supplement: catechin extracts — catechin extracts solution

SUMMARY:
The Purpose of this study is to evaluate the effects of catechin mouth-washing on the removal of intraoral bacteria in the elderly

DETAILED DESCRIPTION:
Catechins are the major components of tea flavonoids and recent in vitro experimental studies have revealed that tea catechin extracts induce bactericidal effects. However, a limited number of studies have been conducted on the clinical effects of tea catechin against bacterial infection and also the effects in the elderly is unclear. Based on these backgrounds, we designed a prospective randomized controlled study to evaluate the effects of catechin mouth washing on oral pathogenic bacterial detected in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* aged over 65 years
* detected oral pathogenic bacterium and revalidated during the wash-out period
* without antibacterial medicine, other mouth-washing remedies during the study
* Obtained written informed consent before participation

Exclusion Criteria:

* possessing some infectious diseases in need of therapy
* possessing tea or catechin allergy
* diagnosed as inadequate for other reasons to participate the study by principal investigator

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Removal of intraoral pathogenic bacteria identified before the study | After intervention

SECONDARY OUTCOMES:
Reduction of intraoral bacteria after the study | After intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamada, MD, PhD, Study Chair — University of Shizuoka
Locations (1):
- White cross nursing home, Higashimurayama, Tokyo, Japan